CLINICAL TRIAL: NCT06251752
Title: Long Term Evaluation of Clinical and Radiologic Results on Femoro-patellar Joint After High Tibial Osteotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HTO-FR
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis; Deformity Knee
Keywords: knee osteotomy; high tibial osteotomy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: cohort 1: lateral closing wedge high tibial osteotomy cohort 2: medial opening wedge high tibial osteotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral closing wedge high tibial osteotomy (Active Comparator)
  Interventions: Diagnostic Test: X-rays: load bearing inferior limbs, lateral knee, axial patella
- Medial opening wedge high tibial osteotomy (Active Comparator)
  Interventions: Diagnostic Test: X-rays: load bearing inferior limbs, lateral knee, axial patella

INTERVENTIONS:
Diagnostic Test: X-rays: load bearing inferior limbs, lateral knee, axial patella — X-rays at 5 years follow-up minimum

SUMMARY:
Osteotomies are among the oldest orthopedic treatments, in use for over 2000 years and still commonly employed. The basic principle involves making a bone cut to allow the realignment of the limb segment affected by deformity. Today, new knowledge and technologies, understanding of bone healing mechanisms, and the introduction of new fixation methods have made osteotomies one of the preferred treatments for early knee arthritis. They serve as an alternative to joint prosthesis implantation in young patients with medium to high functional demand.

Medial knee osteoarthritis is a pathology increasingly prevalent in today's population. The resulting varus deformity leads to a shift in the load axis on the medial tibial plateau. Osteotomy in this context becomes a therapeutic tool capable of restoring the correct mechanical axis of the lower limb and delaying or avoiding the progression of arthritis, thus avoiding the need for joint replacement.

The two most commonly used techniques are the Closing Wedge Lateral High Tibial Osteotomy (LCW-HTO) and the Opening Wedge Medial High Tibial Osteotomy (MOW-HTO), which are high tibial osteotomies in closure with a wedge removal and in opening with a wedge insertion, respectively.

The medium to long-term effects of this procedure, in terms of survival and modification of the tibial slope, have been extensively studied, as evidenced by the extensive literature on the subject. However, the effect of this intervention, in its two variants, on the progression of femoro-patellar arthritis and the height of the patella remains poorly investigated to date.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of medial unicompartmental knee osteoarthritis (Outerbridge III-IV)
2. Follow-up > 60 months
3. Completeness of clinical and radiographic documentation.
4. Previous valgus osteotomy procedure (MOW-HTO or LCW-HTO)
5. Age <65 years

Exclusion Criteria:

1. Patients with previous injuries affecting the involved lower limb.
2. Patients with prior traumatic, septic, and rheumatoid arthritis.
3. Patients with previous alterations of the patellofemoral joint.
4. Patients with knee ligament injuries.
5. Patients with confirmed neuromuscular disorders or psychomotor disturbances.
6. Patients with congenital generalized hypermobility syndrome.
7. Patients with severe pathologies in other organs or systems limiting activities of daily living (ADL).
8. Patients who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
patellar height | baseline time 0
  RX measurement of patellar height
femoral-patellar arthritis | baseline time 0
  RX evaluation of femoral-patellar arthritis

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | baseline time 0
  KOOS assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Kujala score | baseline time 0
  Assessment of patellofemoral disorders: subjective symptoms and functional limitations.
Range of Motion | baseline time 0
  ROM expresses in degrees the degree of range of motion that a joint can perform along its full range of motion whether active or passive through an external aid.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brouwer RW, Huizinga MR, Duivenvoorden T, van Raaij TM, Verhagen AP, Bierma-Zeinstra SM, Verhaar JA. Osteotomy for treating knee osteoarthritis. Cochrane Database Syst Rev. 2014 Dec 13;2014(12):CD004019. doi: 10.1002/14651858.CD004019.pub4. PMID 25503775
- [Result] Coventry MB. Upper tibial osteotomy for osteoarthritis. J Bone Joint Surg Am. 1985 Sep;67(7):1136-40. No abstract available. PMID 4030836
- [Result] Amendola A, Bonasia DE. Results of high tibial osteotomy: review of the literature. Int Orthop. 2010 Feb;34(2):155-60. doi: 10.1007/s00264-009-0889-8. Epub 2009 Oct 17. PMID 19838706